CLINICAL TRIAL: NCT02622113
Title: An Open-Label, Multicenter Study to Evaluate the Long-Term Safety, Tolerability and Efficacy of Canagliflozin (TA-7284) as add-on to Insulin in Subjects With Type 2 Diabetes Mellitus
Brief Title: Long-Term Safety Study of Canagliflozin (TA-7284) in Combination With Insulin in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA-7284-13
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Canagliflozin; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Canagliflozin (TA-7284) ＋insulin (Experimental)
  Interventions: Drug: Canagliflozin (TA-7284); Drug: Insulin

INTERVENTIONS:
Drug: Canagliflozin (TA-7284) — The patients will receive Canagliflozin orally for 36 weeks
Drug: Insulin

SUMMARY:
This extension study was designed to evaluate the safety and efficacy of Canagliflozin (TA-7284) in combination with Insulin in patients with type 2 Diabetes Mellitus. The extension study was an extension to double-blind study of 16 weeks (TA-7284-11)

DETAILED DESCRIPTION:
This is an open-label extension study to evaluate the safety and efficacy of Canagliflozin (TA-7284) in combination with insulin in Japanese patients with Type 2 diabetes mellitus, who are not optimally controlled on diet and exercise. The patients will enroll from the double-blind study of 16 weeks and receive TA-7284 100mg orally for 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients should complete the week 16 assessments in the double-blind study (TA-7284-11)

Exclusion Criteria:

* Patients with hereditary glucose-galactose malabsorption or primary renal glucosuria
* Patients with severe diabetic complications (proliferative diabetic retinopathy, stage 4 nephropathy, or serious diabetic neuropathy)
* Patients with serious renal or hepatic disease
* Patients who are the excessive alcohol addicts
* Patients who are pregnant, lactating and probably pregnant patients and patients who can not agree to contraception

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2014-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation
Locations (7):
- Japan (7):
  - Reserch site, Chugoku
  - Reserch site, Chūbu
  - Reserch site, Hokkaido
  - Reserch site, Kanto
  - Reserch site, Kinki
  - Reserch site, Kyushu
  - Reserch site, Tōhoku

REFERENCES:
- [Result] Inagaki N, Harashima SI, Kaku K, Kondo K, Maruyama N, Otsuka M, Kawaguchi Y, Iijima H. Long-term efficacy and safety of canagliflozin in combination with insulin in Japanese patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2018 Apr;20(4):812-820. doi: 10.1111/dom.13152. Epub 2017 Dec 5. PMID 29110384

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of patients continued treatment in this study after TA-7284-11 study was 139. Four patients in the CANA/CANA group who did not continued this study were included in the analysis set. Analysis of this study was conducted 143 patients.
Groups:
- Placebo/CANA + Insulin: Canagliflozin(CANA) 100mg once daily for 36 weeks, followed placebo for 16 weeks in TA-7284-11 study
- CANA/CANA + Insulin: Canagliflozin(CANA) 100mg once daily for 36 weeks, followed Canagliflozin(CANA) for 16 weeks in TA-7284-11 study
Period: Overall Study
Arm/Group | Placebo/CANA + Insulin | CANA/CANA + Insulin
Started | 67 | 76
Completed | 62 | 66
Not Completed | 5 | 10
Not completed — Adverse Event | 4 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Stopping Criteria | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/CANA + Insulin | CANA/CANA + Insulin | Total
Number analyzed (Participants) | 67 | 76 | 143
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 47 | 93
  >=65 years | 21 | 29 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 32 | 53
  Male | 46 | 44 | 90

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability Assessed by Adverse Events (Number of Participants Experiencing With Adverse Events)
Time Frame: Placebo/CANA: 36 Weeks, CANA/CANA: 52 Weeks
Population: One patient of CANA/CANA group who mistakenly received placebo during TA-7284-11 study, did not continued this study. This patient was included in the full analysis set and was not included in the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/CANA + Insulin | CANA/CANA + Insulin
Number analyzed (Participants) | 67 | 75
Participants
  Serious Adverse Event | 7 | 7
  Adverse Event | 57 | 69

2. Secondary Outcome: Change in Percentage of HbA1c
Time Frame: Placebo/CANA: Baseline, 36 Weeks; CANA/CANA: Baseline, 52 Weeks
Population: Full analysis set, last observation carried forward.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Placebo/CANA + Insulin | CANA/CANA + Insulin
Number analyzed (Participants) | 67 | 76
percentage of HbA1c | -1.09 (0.85) | -0.88 (0.86)

3. Secondary Outcome: Change in Fasting Plasma Glucose
Time Frame: Placebo/CANA: Baseline, 36 Weeks; CANA/CANA: Baseline, 52 Weeks
Population: Full analysis set, last observation carried forward. Outcome measure for two patients of Placebo/CANA group and one patient of CANA/CANA group was not assessed at a certain timepoint due to dropout.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo/CANA + Insulin | CANA/CANA + Insulin
Number analyzed (Participants) | 65 | 75
mg/dL | -33.1 (44.1) | -32.8 (45.7)

4. Secondary Outcome: Percentage Change in Body Weight
Time Frame: Placebo/CANA: Baseline, 36 Weeks; CANA/CANA: Baseline, 52 Weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo/CANA + Insulin | CANA/CANA + Insulin
Number analyzed (Participants) | 65 | 75
percent change | -1.40 (2.54) | -2.14 (2.75)

ADVERSE EVENTS:
Time Frame: Placebo/CANA: 36 Weeks, CANA/CANA: 52 Weeks
Arm/Group | Placebo/CANA + Insulin | CANA/CANA + Insulin
Serious Adverse Events (participants affected / at risk) | 7/67 | 7/75
Other Adverse Events (participants affected / at risk) | 49/67 | 56/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/CANA + Insulin (N=67) | CANA/CANA + Insulin (N=75)
Appendicitis perforated (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Retinal tear (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Alcoholic liver disease (Hepatobiliary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/CANA + Insulin (N=67) | CANA/CANA + Insulin (N=75)
Bronchitis (Infections and infestations) | 4 | 6
Nasopharyngitis (Infections and infestations) | 17 | 26
Pharyngitis (Infections and infestations) | 3 | 6
Upper respiratory tract infection (Infections and infestations) | 3 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 22 | 29
Insomnia (Psychiatric disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 6 | 2
Pollakiuria (Renal and urinary disorders) | 4 | 5
Blood glucose decreased (Investigations) | 16 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other